CLINICAL TRIAL: NCT05083689
Title: Combined Intravitreal Bevacizumab With Topical Timolol-Dorzolamide Eye Drops in Diabetic Macular Edema
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zahra Rabbani Khah, Head of ophthalmic research center, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14002
Record Dates: First submitted 2021-10-06; First posted 2021-10-19 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — Timolol; dorzolamide; Lubricant Eye Drops

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Injections of 1.25 mg of intravitreal bevacizumab with topical drops of Timolol and Dorzolamide (Active Comparator): 31 cases in intervention group receive injections of 1.25 mg of intravitreal bevacizumab monthly for 3 months (months 0, 1 and 2) with topical drops of Timolol twice a day and Dorzolamide twice a day
  Interventions: Drug: Injections of 1.25 mg of intravitreal bevacizumab with Timolol and Dorzolamide
- Injections of 1.25 mg of intravitreal bevacizumab with artificial tears (Placebo Comparator): 31 cases in control group receive intravitreal injection of 1.25 mg bevacizumab monthly for 3 months (months 0, 1 and 2) plus artificial tears (twice a day as a placebo)
  Interventions: Drug: Injections of 1.25 mg of intravitreal bevacizumab with artificial tears

INTERVENTIONS:
Drug: Injections of 1.25 mg of intravitreal bevacizumab with Timolol and Dorzolamide — 31 cases in intervention group receive injections of 1.25 mg of intravitreal bevacizumab monthly for 3 months (months 0, 1 and 2) with topical drops of Timolol twice a day and Dorzolamide twice a day
  Arms: Injections of 1.25 mg of intravitreal bevacizumab with topical drops of Timolol and Dorzolamide
Drug: Injections of 1.25 mg of intravitreal bevacizumab with artificial tears — 31 cases in control group receive intravitreal injection of 1.25 mg bevacizumab monthly for 3 months (months 0, 1 and 2) plus artificial tears (twice a day as a placebo)
  Arms: Injections of 1.25 mg of intravitreal bevacizumab with artificial tears

SUMMARY:
This study is a double-blind randomized clinical trial in Diabetic patients (type 2) over 18 years of age who have diabetic macular edema with involvement of the central 1 millimeter (central macular thickness is more than 300 μm) and BCVA 20/30 or less who visit the retina clinic of Labbafinejad Hospital Are studied. (In patients with bilateral macular edema, only one eye is included in the study.) Complete ocular examinations (including best corrected visual acuity - anterior segment - intraocular pressure - dilated pupil funduscopy with severity of diabetic retinopathy), optical coherence tomography (OCT), EDI-OCT( Enhanced Depth Imaging Optical Coherence Tomography ) - as well as Optical coherence tomography angiography (OCTA ) are performed for all patients at baseline. Blood tests are also taken from patients for fasting blood sugar and HbA1C. Patients are then randomly divided into two groups. The first group is treated with injections of 1.25 mg of intravitreal bevacizumab monthly for 3 months (months 0, 1 and 2) with topical drops of Timolol twice a day and Dorzolamide twice a day. For the second group (control group), 3 injections of 1.25 mg of intravitreal bevacizumab monthly with artificial tears (twice a day as a placebo) are prescribed. Patients in both groups are visited 1 month after the third basic intravitreal bevacizumab (IVB) injection and complete ophthalmology examinations are performed and central thickness of macula is recorded based on the patient's OCT as well as the need for IVB re-injection. EDI (Enhanced Depth Imaging)-OCT and OCTA are performed again for all patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Diabetic Melitus type 2
* Patients with center-involving diabetic macular edema (central macular edema > 300 micrometer)
* Patients have diabetic retinopathy at the stage of nonproliferative diabetic retinopathy (NPDR) or early PDR (proliferative diabetic retinopathy) or regressed PDR
* In patients with bilateral macular edema, only one eye is included in the study.

Exclusion Criteria:

* uncomplicated cataract surgery
* history of cataract surgery during last 4 months
* history of Panretinal Photocoagulation (PRP) during last 4 months
* any retinochoroidal disease except Diabetic retinopathy
* optic disc pathology
* patient with high-risk PDR or advanced PDR
* one-eye patients
* patient with glaucoma or uveitis
* pregnant or lactating patients
* patients whom topical Timolol or Dorzolamide are prohibited for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2021-10-06 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Central macular thickness | 1 month
  Measured by EDI-OCT

SECONDARY OUTCOMES:
Best corrected visual acuity (BCVA) | 1 month
  By ophthalmology resident with subjective and objective refraction

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmic Research Center, Tehran, Iran

REFERENCES:
- [Derived] Fekri S, Rabiei A, Hooshmandi S, Nouri H, Abtahi SH. The effect of combination therapy with intravitreal bevacizumab and topical timolol-dorzolamide eye drops on diabetic macular edema: a double-blind randomized controlled trial. Int Ophthalmol. 2024 Feb 20;44(1):101. doi: 10.1007/s10792-024-03005-z. PMID 38376643